CLINICAL TRIAL: NCT01745757
Title: Cohort Study of Prospective Validation of Predictive Factors and Biological Imaging of Response to Bevacizumab (AVASTIN ®) in Combination With Weekly Paclitaxel Chemotherapy in First Line Treatment Patients With Metastatic Breast Cancer
Brief Title: Cohort Study of Prospective Validation of Predictive Factors and Biological Imaging of Response to Bevacizumab and Paclitaxel in Patients With Metastatic Breast Cancer
Acronym: COMET
Status: Completed | Type: Observational
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Other Study IDs: UC-0102/1203 - GRT02; 2012-A00244-39 (Registry Identifier: ID RCB); GRT02 (Other: UNICANCER)
Record Dates: First submitted 2012-09-18; First posted 2012-12-10 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Metastatic; Breast Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: first line treatment for metastatic breast cancer
  Interventions: Drug: Bevacizumab; Drug: paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Treatments received by patients in this study are prescribed in the context of standard care
Drug: paclitaxel — Treatments received by patients in this study are prescribed in the context of standard care

SUMMARY:
Bevacizumab plus chemotherapy improves response rates and prolongs PFS when used as first- and second-line therapy for advanced breast cancer. However, bevacizumab has not improved OS in the individual studies currently reported. In Europe, EMA has maintained its indication associated with weekly paclitaxel in first line metastatic breast cancer and more recently with capecitabine based on RIBBON 1 trial's results.

The identification of patient subsets that receive the most clinical benefit would enable more specific treatment administration of bevacizumab and allow patients unlikely to benefit the opportunity to seek other treatment modalities. Unfortunately, despite efforts to identify patient subsets with a differential benefit from bevacizumab, no validated biomarkers have been defined.

The Avastin cohort is a unique opportunity to investigate various biological and imaging parameters which could be related to clinical benefit of the combination of bevacizumab and weekly paclitaxel in first line metastatic breast cancer in a homogeneously treated population in French cancer centers. This trial will gather the expertise of several translational research platforms of different cancer centers from the UNICANCER consortium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old.
* Histologically confirmed breast adenocarcinoma, metastatic (measurable or unmeasurable lesion), HER2 negative (on the last tumor tissue analyzed), Patient to receive first-line chemotherapy paclitaxel and bevacizumab in a weekly manner as recommended by the EMEA.
* Hormone receptor status known
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy ≥12 weeks.
* Women of childbearing age (except amenorrhea of at least 24 months) must have a negative pregnancy test serum within 28 days before starting treatment. In the absence of serum test, a urine pregnancy test (within 7 days before the first dose of bevacizumab) is required.
* Informed consent form duly signed and dated by patient

Exclusion Criteria:

* Prior chemotherapy for metastatic disease ;
* Concomitant hormone therapy
* The patient must not have undergone radiation therapy for the treatment of metastatic disease (except cases of analgesic radiotherapy for bone pain due to metastases).
* Pregnant or nursing woman or woman of childbearing age (except amenorrhea for at least 24 months) who does not use an effective nonhormonal contraceptive method (intrauterine device, barrier method associated with the use of a spermicidal gel or surgical castration) for the duration of the study and 6 months after paclitaxel administration and / or bevacizumab.
* Man who does not accept to use effective contraception during the study period and 6 months after paclitaxel administration and / or bevacizumab.
* Known hypersensitivity to paclitaxel and / or to bevacizumab or to any excipients.
* Patient unable to undergo medical test for geographical, social or psychological reasons.
* Patient deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2012-06; Primary Completion 2022-06 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Measure of the initial rates and changes in CEC / CLC (Biological study) and measure of the visceral fat (imaging study) as predictors of progression-free survival (PFS) and response to bevacizumab and paclitaxel | 2 years

SECONDARY OUTCOMES:
Identification of new biomarkers as predictive factors of progression free survival (PFS), overall survival (OS) and of response to bevacizumab and paclitaxel. | 2 years
  These biomarkers will be selected from biological studies, proteomics and pharmacogenetics.
Quality of Life assessment | 2 years
The Biomarkers selected from our biological, proteomic and pharmacogenetic studies will be correlated to the safety. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves PIERGA, MD, PhD, Principal Investigator — Institut Curie Paris
Locations (19):
- France (19):
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - CHU Grenoble, Grenoble
  - Centre Leon Berard, Lyon
  - Hôpital Européen, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Hospitalier, Roanne
  - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Result] Bortolini Silveira A, Bidard FC, Tanguy ML, Girard E, Tredan O, Dubot C, Jacot W, Goncalves A, Debled M, Levy C, Ferrero JM, Jouannaud C, Rios M, Mouret-Reynier MA, Dalenc F, Hego C, Rampanou A, Albaud B, Baulande S, Berger F, Lemonnier J, Renault S, Desmoulins I, Proudhon C, Pierga JY. Multimodal liquid biopsy for early monitoring and outcome prediction of chemotherapy in metastatic breast cancer. NPJ Breast Cancer. 2021 Sep 9;7(1):115. doi: 10.1038/s41523-021-00319-4. PMID 34504096
- [Result] Gal J, Milano G, Brest P, Ebran N, Gilhodes J, Llorca L, Dubot C, Romieu G, Desmoulins I, Brain E, Goncalves A, Ferrero JM, Cottu PH, Debled M, Tredan O, Chamorey E, Merlano MC, Lemonnier J, Etienne-Grimaldi MC, Pierga JY. VEGF-Related Germinal Polymorphisms May Identify a Subgroup of Breast Cancer Patients with Favorable Outcome under Bevacizumab-Based Therapy-A Message from COMET, a French Unicancer Multicentric Study. Pharmaceuticals (Basel). 2020 Nov 23;13(11):414. doi: 10.3390/ph13110414. PMID 33238394
- [Result] Vasseur A, Cabel L, Tredan O, Chevrier M, Dubot C, Lorgis V, Jacot W, Goncalves A, Debled M, Levy C, Ferrero JM, Jouannaud C, Luporsi E, Mouret-Reynier MA, Dalenc F, Lemonnier J, Savignoni A, Tanguy ML, Bidard FC, Pierga JY. Prognostic value of CEC count in HER2-negative metastatic breast cancer patients treated with bevacizumab and chemotherapy: a prospective validation study (UCBG COMET). Angiogenesis. 2020 May;23(2):193-202. doi: 10.1007/s10456-019-09697-7. Epub 2019 Nov 26. PMID 31773439